CLINICAL TRIAL: NCT03809195
Title: Clinical Hypnosis in Pediatric Crohn's Disease
Acronym: HypnoCrohns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Amanda Lee, Clinical Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 181436
Record Dates: First submitted 2019-01-03; First posted 2019-01-18 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pediatric Crohns Disease
Keywords: hypnosis; inflammatory bowel disease; mind-body; brain-gut; hypnotherapy; quality of life; psychosocial
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: intervention group versus control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis Intervention (Experimental): The intervention is clinical hypnosis--a single in-person session followed by instructions to listen to audio recordings at home. The sessions consist of the provider's voice guiding the participant into a relaxed and focused state and providing therapeutic suggestions--for example, to replace discomfort with a more pleasant sensation, to ease anxiety, and to increase energy.
  Interventions: Behavioral: Clinical Hypnosis
- Waitlist Control (No Intervention): This group will serve as a control comparison and be offered the intervention after control data collection is complete.

INTERVENTIONS:
Behavioral: Clinical Hypnosis — See information in arm/group description. Four different audio recordings are provided electronically, each approximately 20 minutes in length. Participants are encouraged to listen to one daily.
  Arms: Hypnosis Intervention

SUMMARY:
Inflammatory bowel disease (IBD), which includes Crohn's disease (CD) and ulcerative colitis (UC), is a chronic, immune-mediated disease increasingly prevalent in youth. Patients with IBD experience pain, fatigue, altered bowel habits, psychological distress, and reduced quality of life. Regardless of disease activity, persistent pain and psychiatric comorbidities both have a negative impact on quality of life. Alongside standard pharmacologic and nutritional therapies, clinical hypnosis is a complementary therapy that may improve physical and psychosocial outcomes in these patients. Clinical hypnosis consists of guiding the patient into a relaxed and focused state and providing therapeutic suggestions to induce desired physiologic and psychologic change. Children and adolescents are excellent candidates for hypnosis by virtue of their vivid imaginations. Hypnosis is effective in management of functional abdominal pain, irritable bowel syndrome, anxiety, chronic pain, and distress related to medical procedures. To date, there are no clinical trials that evaluate the effects of hypnosis in pediatric patients with IBD, but there is strong conceptual support for its role in improving pain and psychological distress in these patients. In addition to genetic, environmental, and microbial influences, a growing body of evidence supports the role of a dysregulated brain-gut axis and chronic stress in IBD. Animal and human studies demonstrate the effect of stress on the immune system and gastrointestinal tract. Studies show that the benefits of hypnosis may extend to its role in increasing vagal tone and regulating the immune system via the brain-gut axis. Adults with UC receiving a hypnosis intervention demonstrated improved remission and decreased inflammatory markers. Case series suggest that children with inflammatory bowel disease benefit from hypnosis, and it can be safely and easily delivered via audio recordings. Patients with IBD are interested in integrative therapies to reduce symptoms and improve quality of life, and a biopsychosocial approach is essential in their care. The addition of hypnosis may improve outcomes through influence on stress, inflammation, coping, symptom perception, and quality of life.

The investigators hypothesize that pediatric patients with CD participating in a clinical hypnosis intervention as an adjunct to standard of care will report improved quality of life compared to a waitlist control group. The specific aims of the study are as follows: (1) To implement hypnosis as an adjunctive therapy in adolescents with CD. (2) To evaluate the impact of hypnosis in CD on measures of quality of life. (3) To evaluate the impact of hypnosis in CD on pain, depression, anxiety, sleep, and coping.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Crohn's disease at least 3 months prior to enrollment
* Inactive, mild, or moderate disease activity by Improve Care Now Physician's Global Assessment (ICN PGA) at most recent GI clinic visit
* Ages 12-18 years at time of enrollment
* English-speaking and with the normal cognitive development required to understand the verbal instructions/suggestions provided in the hypnosis session/audio recordings and to understand and complete the written surveys
* Has daily access to an electronic device (ex. smartphone, computer) that can receive text messages or e-mail, on which online surveys can be completed, and on which the participant can access and listen to audio recordings.

Exclusion Criteria:

* Patients diagnosed with Crohn's disease less than 3 months prior to enrollment
* Severe disease activity per ICN PGA at most recent GI clinic visit
* Age < 12 years or > 18 years
* Non-English speaking or having a cognitive disability that precludes understanding the verbal instructions/suggestions provided in the hypnosis session/audio recordings and the completion of written surveys
* Lacks daily access to an electronic device (ex. smartphone, computer) that can receive text messages or e-mail, on which online surveys can be completed, and on which the participant can access and listen to audio recordings.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
IMPACT-III | Change from baseline to 8 weeks.
  Pediatric inflammatory bowel disease-specific health-related quality of life measure. "IMPACT" is not an abbreviation, but rather the name of the scale. Minimum score 0 to maximum score 100, with higher signifying better quality of life. Subjects get a total score (0 to 100) and a score for each of six subscales (0 to 100): Bowel Symptoms (7 items), Treatment/Interventions (3 items), Social Functioning (12 items), Emotional Functioning (7 items), Body Image (3 items), Systemic Symptoms (3 items). Each of the 35 total items has five multiple choice options and is given a score of 0, 25, 50, 75, or 100 points. The subscale scores are an average of the scores for each item that corresponds to that subscale. The total score is an average of all item scores.
Modified Cantril Ladder | Change from baseline to 8 weeks.
  Single item quality of life measure. From 0 to 10, with 10 representing the best quality of life.
PedsQL 4.0 Generic Core Scale, Parent Proxy | Change from baseline to 8 weeks.
  "PedsQL" refers to Pediatric Quality of Life. This is a pediatric 23-item measure of health-related quality of life. Questions fall under one of five domains: Physical Functioning (8 items), Emotional Functioning (5), Social Functioning (5 items), School Functioning (5 items). Yields a total score and two summary scores-Physical Health (comprised of physical functioning domain) and Psychosocial Health (comprised of each item in the 5-item emotional, social, and school functioning domains). Each item is rated on a 5-point Likert scale. Total score and the two summary scores are linearly transformed into a 0 to 100 point scale, with higher scores representing better quality of life.

SECONDARY OUTCOMES:
PROMIS Pediatric Anxiety, short form | Change from baseline to 8 weeks.
  PROMIS stands for Patient-Reported Outcomes Measurement Information System. This measure is 8 items each scored from 1 to 5 points, with the lowest possible raw score being 8 and the highest possible raw score being 40. Higher scores indicate greater anxiety, i.e. worse. The raw score is translated into a T-score. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
PROMIS Pediatric Depressive Symptoms, short form | Change from baseline to 8 weeks.
  PROMIS stands for Patient-Reported Outcomes Measurement Information System. This measure is 8 items each scored from 1 to 5 points, with the lowest possible raw score being 8 and the highest possible raw score being 40. Higher scores indicate greater depressive symptoms, i.e. worse. The raw score is translated into a T-score. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
PROMIS Pediatric Sleep Disturbance, short form | Change from baseline to 8 weeks.
  PROMIS stands for Patient-Reported Outcomes Measurement Information System. This measure is 8 items each scored from 1 to 5 points, with the lowest possible raw score being 8 and the highest possible raw score being 40. Higher scores indicate greater sleep disturbance, i.e. worse sleep. The raw score is translated into a T-score. The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
Pain Beliefs Questionnaire, short form | Change from baseline to 8 weeks.
  This is an 18-item measure designed assess youth's beliefs about their abdominal pain. It is comprised of three subscales each with 6 items-Pain Threat, Problem-Focused Coping Efficacy (PFCE), and Emotion-Focused Coping Efficacy (EFCE). The respondent rates each item on how true the statement is for them on a 5-point scale ranging from 0 ("not at all true") to 4 ("very true"). Subscale scores are computed by averaging the items pertaining to each subscale. For Pain Threat, higher score indicates stronger beliefs that one's pain represents a personal threat. For the PFCE and EFCE subscales, higher scores indicate a stronger belief in one's ability to cope with pain.
Abdominal Pain Intensity | Change from baseline to 8 weeks.
  Two items combined for a total score, range from 0 to 20, with higher scores representing greater pain intensity. Each item rated on a scale from 0 (no pain) to 10 (most possible pain). The first item assesses the respondent's worst pain in the past week, and the second item assesses the usual intensity of the pain experienced during the past week. Adapted from the Abdominal Pain Index, with permission.
Healthcare utilization | Change from baseline to 8 weeks.
  By parent report, total number of contacts health care provider for their child in the past 8 weeks, other than previously scheduled check-ups, including emergency department visits, urgent care visits, and phone calls or messages to the doctor's office
School absences | Change from baseline to 8 weeks.
  By parent report, number of days of school the child has missed in the past 8 weeks (choices: 0, 1-3, 4-6, 7-10, more than 10 days). If on school break, parent asked to estimate as if school was in session--for example, how many days the child had to miss usual activities.
Abdominal Pain Frequency | Change from baseline to 8 weeks.
  How many days did the respondent experience pain in the past week, with options being never, 1-2 days, 3-4 days, 5-6 days, or daily, with greater frequency of pain being worse. Adapted from the Abdominal Pain Index, with permission.

OTHER OUTCOMES:
IMPACT-III | Change from baseline to secondary time point at 16 weeks.
  Pediatric inflammatory bowel disease-specific health-related quality of life measure. "IMPACT" is not an abbreviation, but rather the name of the scale. Minimum score 0 to maximum score 100, with higher signifying better quality of life. Subjects get a total score (0 to 100) and a score for each of six subscales (0 to 100): Bowel Symptoms (7 items), Treatment/Interventions (3 items), Social Functioning (12 items), Emotional Functioning (7 items), Body Image (3 items), Systemic Symptoms (3 items). Each of the 35 total items has five multiple choice options and is given a score of 0, 25, 50, 75, or 100 points. The subscale scores are an average of the scores for each item that corresponds to that subscale. The total score is an average of all item scores.
PedsQL 4.0 Generic Core Scale, Parent Proxy | Change from baseline to secondary time point at 16 weeks.
  "PedsQL" refers to Pediatric Quality of Life. This is a pediatric 23-item measure of health-related quality of life. Questions fall under one of five domains: Physical Functioning (8 items), Emotional Functioning (5), Social Functioning (5 items), School Functioning (5 items). Yields a total score and two summary scores-Physical Health (comprised of physical functioning domain) and Psychosocial Health (comprised of each item in the 5-item emotional, social, and school functioning domains). Each item is rated on a 5-point Likert scale. Total score and the two summary scores are linearly transformed into a 0 to 100 point scale, with higher scores representing better quality of life.
Modified Cantril Ladder | change over time monitored weekly for 8 weeks then at secondary time point at 16 weeks
  Single item quality of life measure. From 0 to 10, with 10 representing the best quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda D Lee, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone AL, Walker LS, Laird KT, Shirkey KC, Smith CA. Pediatric Pain Beliefs Questionnaire: Psychometric Properties of the Short Form. J Pain. 2016 Sep;17(9):1036-44. doi: 10.1016/j.jpain.2016.06.006. Epub 2016 Jun 27. PMID 27363626
- [Background] Forrest CB, Meltzer LJ, Marcus CL, de la Motte A, Kratchman A, Buysse DJ, Pilkonis PA, Becker BD, Bevans KB. Development and validation of the PROMIS Pediatric Sleep Disturbance and Sleep-Related Impairment item banks. Sleep. 2018 Jun 1;41(6). doi: 10.1093/sleep/zsy054. PMID 29546286
- [Background] Zhang YZ, Li YY. Inflammatory bowel disease: pathogenesis. World J Gastroenterol. 2014 Jan 7;20(1):91-9. doi: 10.3748/wjg.v20.i1.91. PMID 24415861
- [Background] Mackner LM, Greenley RN, Szigethy E, Herzer M, Deer K, Hommel KA. Psychosocial issues in pediatric inflammatory bowel disease: report of the North American Society for Pediatric Gastroenterology, Hepatology, and Nutrition. J Pediatr Gastroenterol Nutr. 2013 Apr;56(4):449-58. doi: 10.1097/MPG.0b013e3182841263. PMID 23287808
- [Background] Kunz JH, Hommel KA, Greenley RN. Health-related quality of life of youth with inflammatory bowel disease: a comparison with published data using the PedsQL 4.0 generic core scales. Inflamm Bowel Dis. 2010 Jun;16(6):939-46. doi: 10.1002/ibd.21128. PMID 19998462
- [Background] Vlieger AM, Menko-Frankenhuis C, Wolfkamp SC, Tromp E, Benninga MA. Hypnotherapy for children with functional abdominal pain or irritable bowel syndrome: a randomized controlled trial. Gastroenterology. 2007 Nov;133(5):1430-6. doi: 10.1053/j.gastro.2007.08.072. Epub 2007 Sep 2. PMID 17919634
- [Background] Palsson OS. Hypnosis Treatment of Gastrointestinal Disorders: A Comprehensive Review of the Empirical Evidence. Am J Clin Hypn. 2015 Oct;58(2):134-58. doi: 10.1080/00029157.2015.1039114. PMID 26264539
- [Background] Bonaz BL, Bernstein CN. Brain-gut interactions in inflammatory bowel disease. Gastroenterology. 2013 Jan;144(1):36-49. doi: 10.1053/j.gastro.2012.10.003. Epub 2012 Oct 12. PMID 23063970
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391